CLINICAL TRIAL: NCT03478371
Title: In-use Randomized, Cross-over, Controlled Double-blind Study of Four Different Tampons
Brief Title: In-use Study of Four Different Tampons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CSD 2017-164
Record Dates: First submitted 2018-02-05; First posted 2018-03-27 (Actual); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Menstruation
Keywords: tampon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Marketed Tampon D (Sham Comparator): Regular absorbency tampon
  Interventions: Device: tampon D
- Marketed Tampon M (Sham Comparator): Regular absorbency tampon
  Interventions: Device: tampon M
- Marketed Tampon T (Sham Comparator): Regular absorbency tampon
  Interventions: Device: tampon T
- Marketed Tampon V (Sham Comparator): Regular absorbency tampon
  Interventions: Device: tampon V

INTERVENTIONS:
Device: tampon D — regular absorbency tampon
  Arms: Marketed Tampon D
Device: tampon M — regular absorbency tampon
  Arms: Marketed Tampon M
Device: tampon T — regular absorbency tampon
  Arms: Marketed Tampon T
Device: tampon V — regular absorbency tampon
  Arms: Marketed Tampon V

SUMMARY:
This study will evaluate the impact on vaginal health of four different tampons using gynecologic assessment and subjective assessment of comfort during in-use conditions

ELIGIBILITY:
Inclusion Criteria: To be considered eligible for enrollment into this study subjects must meet the following criteria:

1. signed the Informed Consent;
2. female, between 18 and 55 years of age;
3. agree to practice abstinence or use an effective form of birth control (e.g. intrauterine device, oral contraceptives, contraceptive implants or injections, diaphragm with spermicide, cervical cap, or constant use of condom) for at least the past 4 months and willing to continue throughout the study or have had a tubal ligation or your partner has had a vasectomy at least 4 months before being enrolled in the study;
4. be in generally good health without clinically significant disease as determined by investigator or designee based on medical history and vaginal exam;
5. for at least the last 4 months, have a consistent menstrual cycle lasting 21-35 days with menstrual bleeding lasting at least 3 days' duration;
6. primarily use tampons for their feminine protection needs during their periods (may use provided pads and/or pantiliners as back-up to tampon);
7. typically use Regular (6-9 grams) absorbency tampons for the majority of their period,
8. wears tampons during menstruation with no history of abnormal discomfort;
9. last pap smear was normal in the past 3 years or a normal pap with a negative HPV in the past 5 years (age 18-21 does NOT need a PAP if they have never been sexually active), per standard of care (per ACOG guidelines), (self-reported);
10. agree to refrain from vaginal intercourse within 48 hours of each vaginal exam scheduled visit;
11. agree to refrain from showering within twelve (12) hours or bathing within twenty-four (24) hours (1 day) of each visit (except Visit 2);
12. agree to refrain from using douching substances, feminine hygiene products, and to not apply powders, perfumes, wipes, lotions, creams, or emollients to their genital area 48 hours prior to the screening visit and through the completion of the study, if accepted to participate in the study;
13. agree to refrain from taking anti-inflammatory, antihistamine and/or, steroid systemic and/or topical, (including new hormonal contraceptives) medications until they have completed the study (e.g. Advil, Motrin, Benadryl, etc.);
14. agree to only use the tampons, pads and pantiliners supplied at each study visit for her menstrual protection while participating in this study;
15. be willing and able to comply with the study requirements;
16. agree to complete all study questionnaires;
17. agree to refrain from participation in other concurrent clinical research studies;
18. agree to refrain from genital hair removal (e.g. waxing/shaving, etc.) while on the study;
19. agree to refrain from using antibacterial body soap while on the study (e.g. Safeguard)

Exclusion Criteria: Subjects will be excluded from the study if they meet any of the following criteria:

1. have a menstrual abnormality with in the last 4 months (such as oligomenorrhea or amenorrhea);
2. has had a vaginal delivery in the last 6 months;
3. had vaginal surgery, perineal surgery, uterine surgery, miscarriage or abortion in the last 6 months;
4. are pregnant (per urine pregnancy test at screening), or intend to become pregnant in the next 5 months;
5. have a history of Toxic Shock Syndrome (TSS);
6. have a history of heart valve replacement;
7. have had an abnormal Pap in either of your last 2 Pap Smears;
8. have taken steroids (systemic and/or topical), corticosteroids, antihistamines, and/or anti-inflammatories within the past seven days (excludes hormonal contraception);
9. have a history of immunosuppressive drug therapy, chemotherapy, or radiation therapy;
10. have uncontrolled and/or unstable diabetes (exception...stable dose of Diabetic medication for at least 6 months prior to enrollment) in the opinion of the Investigator;
11. have a vulvar piercing;
12. have a history of genital herpes;
13. within the last 6 months have had endometrial disease/uterine fibroids with symptoms of heavy menstrual flow (super plus tampon absorbency use) and/or severe menstrual cramping;
14. have you been diagnosed with a current medical condition which might compromise the immune system functions; including cancer, anemia, leukopenia, leukocyte function deficiency, malnutrition, or chemical dependence (e.g. opiates, marijuana etc.) (self-reported);
15. have clinically diagnosed genital warts, lesions, and/or vaginal infections (such as bacterial vaginosis (BV), Candida spp., Trichomonas vaginalis) at the screening visit;
16. have clinically diagnosed active or vaginal infections (Chlamydia trachomatis and/or Neisseria gonorrhoeae) identified through lab results from the microbiological sample obtained at the screening visit;
17. has urinary incontinence which causes subject to regularly use and saturate diapers or absorbent panties or pads more than 3 times a week over the last 4 months, or currently under treatment for a pelvic floor disorder (i.e., perineal floor re-education with vaginal probe within last 6 months);
18. have history of or current diagnosis of AIDS/HIV, organ transplant, neoplasia, liver disease, renal disease, deep vein thrombosis, pulmonary embolism, haemophilia, neutropenia, autoimmune disease, major depression or any other medical condition, which in the opinion of the Investigator would preclude study participation (exception...stable dose of Thyroid medication for at least 6 months prior to enrollment);
19. having a vaginal probiotic therapy (self-reported)
20. have participated in a clinical study with exposure to any investigational drug product within 30 days prior to this study;
21. have a vaginal erythema grade of ≥2.0 and/or the presence of abrasions and/or ulcerations as determined by investigator, at the screening visit;
22. have taken antibiotics or antifungals within last 4 weeks (Topical use of antibiotics or antifungals outside the perineal/genitourinary area is allowed at the discretion of the Investigator);
23. have started a new hormonal birth control in the previous 4 months or plan changing hormonal birth control throughout the study period;
24. currently experiencing bladder, uterine or rectal prolapse (investigator to verify at screening visit).
25. history of led or laser vaginal therapy within last 6 months (self-reported)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Noss, MD, Principal Investigator — Site Medical Director
Locations (1):
- Synexus-US, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hochwalt AE, Abbinante-Nissen JM, Bohman LC, Hattersley AM, Hu P, Streicher-Scott JL, Teufel AG, Woeller KE. The safety assessment of tampons: illustration of a comprehensive approach for four different products. Front Reprod Health. 2023 Jun 20;5:1167868. doi: 10.3389/frph.2023.1167868. eCollection 2023. PMID 37408999

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: This was a single center, double-blind 4 treatment, 4 period cross-over design. Each participant received each test product for one menstrual cycle.
Period: Overall Study
Arm/Group | Overall Study
Started | 94
Received Tampon D | 91
Received Tampon M | 92
Recived Tampon T | 90
Received Tampon V | 91
Completed | 89
Not Completed | 5
Not completed — non-compliance | 1
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 94
Age, Continuous [Mean (Full Range); unit: years] | 33.4 [18 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 2
  Asian Indian | 0
  Asian Oriental | 2
  Black | 36
  Caucasian | 51
  Mutli-racial | 0
  Native Hawaiian or Pacific Islander | 0
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Tolerance of Tampon Wear Via Physician Assessment of Vaginal Health
Description: The physician examiner determined tampon tolerance based on the following: 1) Vaginal erythema (0-4 scale), 2) vaginal lacerations (presence or absence), 3) vaginal abrasions (presence or absence), 4) vaginal pH, 5) vaginal discharge
Time Frame: within 72 hours last tampon use
Population: ITT population was the primary population of analysis. The ITT population was defined as those participants who were randomized, received at least one test product and had at least one post-product use measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | Marketed Tampon D | Marketed Tampon M | Marketed Tampon T | Marketed Tampon V
Number analyzed (Participants) | 91 | 92 | 90 | 91
Participants
  Erythema score greater than 0 | 0 | 0 | 0 | 0
  Presence of Ulcerations | 0 | 0 | 0 | 0
  Presence of Abrasions | 0 | 0 | 0 | 0
  Abnormal Vaginal Discharge | 0 | 0 | 0 | 0

2. Primary Outcome: Vaginal pH
Description: Vaginal pH
Time Frame: within 72 hours last tampon use
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pH
Arm/Group | Marketed Tampon D | Marketed Tampon M | Marketed Tampon T | Marketed Tampon V
Number analyzed (Participants) | 91 | 92 | 90 | 91
pH | 4.43 (0.053) | 4.46 (0.061) | 4.40 (0.055) | 4.44 (0.061)

3. Secondary Outcome: Subject Comfort Diary
Description: Diary assessment of tampon wear comfort. This assessment uses a 5-point scale which was summarized using the mean as the summary statistic. This questionnaire measured overall comfort using a +2 to -2 scale that was converted to a 0 to 100 scale: 100 = excellent rating and 0 =poor rating
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Marketed Tampon D | Marketed Tampon M | Marketed Tampon T | Marketed Tampon V
Number analyzed (Participants) | 91 | 92 | 90 | 91
units on a scale | 81.7 (2.60) | 78.5 (2.56) | 74.0 (2.58) | 73.2 (2.57)

4. Secondary Outcome: Subject Comfort Questionnaire
Description: Post-menstruation assessment of tampon wear comfort. This assessment uses a 5-point scale which was summarized using the mean as the summary statistic. This questionnaire measured overall satisfaction using a +2 to -2 scale that was converted to a 0 to 100 scale: 100 = excellent rating and 0 = poor rating
Time Frame: 4 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Marketed Tampon D | Marketed Tampon M | Marketed Tampon T | Marketed Tampon V
Number analyzed (Participants) | 91 | 92 | 90 | 91
units on a scale | 78.4 (3.17) | 71.5 (3.17) | 66.5 (3.17) | 60.9 (3.15)

ADVERSE EVENTS:
Time Frame: six months
Arm/Group | Marketed Tampon D | Marketed Tampon M | Marketed Tampon T | Marketed Tampon V
All-Cause Mortality (participants affected / at risk) | 0/91 | 0/92 | 0/90 | 0/91
Serious Adverse Events (participants affected / at risk) | 1/91 | 0/92 | 0/90 | 0/91
Other Adverse Events (participants affected / at risk) | 0/91 | 0/92 | 0/90 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Marketed Tampon D (N=91) | Marketed Tampon M (N=92) | Marketed Tampon T (N=90) | Marketed Tampon V (N=91)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/71/NCT03478371/Prot_SAP_000.pdf